CLINICAL TRIAL: NCT05053061
Title: Does Pulmonary Rehabilitation With Telerehabilitation Increase Physical Capacity in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Telerehabilitation in COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Cenk Kirakli, M.D., Professor Doctor, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IGHCEAH-ICU6
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: COPD
Keywords: COPD; Pulmonary Rehabilitation; Telerehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation Arm (Experimental)
  Interventions: Behavioral: Application program for pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Application program for pulmonary rehabilitation — Exercise videos for pulmonary rehabilitation

SUMMARY:
The prevalence of chronic obstructive pulmonary disease (COPD) in Turkey is 10%. Patients with COPD have a decreased physical capacity. Decreased physical activity in COPD patients causes an increase in all-cause mortality. Pulmonary rehabilitation contributes to increasing physical capacity and quality of life in COPD patients. However, a limited number of patients have access to pulmonary rehabilitation. Some of the patients drop out of pulmonary rehabilitation due to reasons such as transport difficulties, low social support, and low professional support. In addition, disruption of daily routine is one of the important reasons for this situation. Telerehabilitation can enable more patients to access pulmonary rehabilitation. Education and exercise programs can be followed with telerehabilitation in patients with COPD. An increase in exercise capacity and a decrease in dyspnea have been achieved with telerehabilitation in COPD patients.

Different technologies such as telephone, video conferencing or web sites can be used for telerehabilitation. Also, mobile phone was used to telerehabilitation. To make pulmonary telerehabilitation completely patient-based, we have developed an application suitable for smartphones. The application contains videos which showing how to perform pulmonary rehabilitation exercise videos, and it allows the participants to follow up compliance with pulmonary rehabilitation daily. The application will be downloaded to the smartphones of the participants, and it will be shown how to use the application. Participants will not be shown pulmonary rehabilitation exercises.

This study aims to evaluate the effectiveness of telerehabilitation with the application program on physical capacity, quality of life, and dyspnea perception in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Being diagnosed with COPD
* Not have previously participated in pulmonary rehabilitation
* To able to use smartphone

Exclusion Criteria:

* Under age 18
* Pregnancy
* Have previously participated in pulmonary rehabilitation
* Having any malignacy
* Having any disorder that limit exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
6-min walk test (6MWT) | 8 weeks
  exercise capacity

SECONDARY OUTCOMES:
Short Form-36 (SF-36) | 8 weeks
  Quality of life
St George's Respiratory Questionnaire | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 1University of Health Sciences Turkey, Dr Suat Seren Chest Diseases and Chest Surgery Training and Research Hospital, Intensive Care Unit, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No